CLINICAL TRIAL: NCT04989517
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1b Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of AT193 in the Treatment of Patients With Hidradenitis Suppurativa
Brief Title: Study of Efficacy and Safety of Investigational Treatment in Patients With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azora Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Azora Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS01
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT193 (Experimental): Topical applied daily
  Interventions: Drug: AT193
- Placebo (Placebo Comparator): Topical applied daily
  Interventions: Drug: AT193

INTERVENTIONS:
Drug: AT193 — Topical

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group phase 1b study to evaluate AT193 in approximately 44 participants with HS. The treatment period will be 8 weeks followed by a 2-week nontreatment follow-up. The primary objective of this study is to evaluate the safety and tolerability of AT193. The secondary objectives of this study are to evaluate the preliminary efficacy in the treatment of HS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS or signs and symptoms consistent with HS for at least 3 months before screening in the judgment of the investigator.
* Stable disease for at least 2 months before screening in the judgment of the investigator.
* A woman of childbearing potential must use appropriate contraceptive measures during the study period.
* A woman of childbearing potential must have a negative urine pregnancy test result at screening.
* Written informed consent must be obtained before any study procedure is performed.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Any active skin disease that may interfere with evaluation of study drug or outcome assessment.
* History or evidence of a clinically significant disorder, condition, or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion in the judgment of the investigator.
* Change in smoking or marijuana history within 3 months before Day 1 or planned during study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 10 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - Premier Specialists, Kogarah, New South Wales
  - Novatrials, Kotara, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - North Eastern Health Specialists, Campbelltown, South Australia

IPD SHARING:
Plan to Share IPD: No